CLINICAL TRIAL: NCT01634308
Title: Efficacy and Safety of Bongros-BMP Compared to Bio-oss for Regeneration of Alveolar Bone Tissue After Maxillary Sinus Floor Augmentation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Collaborators: Bio-alpha Co. LTD. (Unknown)
Responsible Party: Sponsor
Other Study IDs: BA05-CP01
Record Dates: First submitted 2012-07-03; First posted 2012-07-06 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Regeneration of Alveolar Tissue After Maxillary Sinus Floor Augmentation
MeSH Terms: interventions — Bio-Oss

ARMS (2):
- Novosis(bongros/BMP-2) (Experimental)
  Interventions: Drug: Novosis(bongros/BMP-2)
- Bio-oss (Active Comparator)
  Interventions: Drug: Bio-oss

INTERVENTIONS:
Drug: Novosis(bongros/BMP-2)
  Arms: Novosis(bongros/BMP-2)
Drug: Bio-oss
  Arms: Bio-oss

SUMMARY:
The purpose of this Clinical study was to evaluate the Efficacy and Safety of bongros-BMP compared to Bio-oss for Regeneration of alveolar bone tissue after Maxillary sinus floor augmentation.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2010-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Oral and Maxillofacial Surgery and School of Dentistry, Seoul National University, Seoul, South Korea

REFERENCES:
- [Derived] Kim HJ, Chung JH, Shin SY, Shin SI, Kye SB, Kim NK, Kwon TG, Paeng JY, Kim JW, Oh OH, Kook MS, Yang HJ, Hwang SJ. Efficacy of rhBMP-2/Hydroxyapatite on Sinus Floor Augmentation: A Multicenter, Randomized Controlled Clinical Trial. J Dent Res. 2015 Sep;94(9 Suppl):158S-65S. doi: 10.1177/0022034515594573. Epub 2015 Jul 16. PMID 26185033